CLINICAL TRIAL: NCT00228839
Title: A Pediatric Phase I Pharmacokinetic Study Using Anti Tumor Necrosis Factor Antibody (Infliximab) for Treatment of Acute Graft Versus Host Disease
Brief Title: GVH 022P: Study Using Anti Tumor Necrosis Factor Antibody (Infliximab) for Treatment of Acute Graft Versus Host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 540-2003
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2007-12

CONDITIONS: Graft vs Host Disease
Keywords: Recipients of an allogeneic hematopoietic stem cell transplant who have acute GVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
Acute graft versus host disease (GVHD) remains one of the most significant and potentially lethal complications of allogeneic bone marrow transplantation. Depending upon the type of transplant, the incidence of acute GVHD varies between 20 - 50% in related donor transplants, or as high as 70 - 90% in unrelated donor transplants. Acute GVHD affects the skin, liver and gastrointestinal (GI) tract and usually occurs within 20 - 40 days of the bone marrow infusion.

Steroids are the standard initial treatment of acute GVHD, with approximately 50% of the patients either free of disease or requiring no further therapy. In the remaining patients, the GVHD either does not respond or it comes back during the tapering of steroids. These patients have a much worse prognosis with a mortality rate greater than 70%. Studies using additional agents such as antithymocyte globulin (ATG), monoclonal antibodies, and anti-lymphocyte globulin showed no improvement over the use of steroids alone. This leads the investigators to look for new immunosuppressive agents that can reduce the risk and severity of acute GVHD.

The major purpose of this study is to evaluate the way the body uses and absorbs (the pharmacokinetic profile) a drug called anti tumor necrosis factor antibody (infliximab) for the treatment of acute GVHD. Infliximab is currently indicated for the treatment of immunologic-based diseases (rheumatoid arthritis, moderately to severely active Crohn's disease, and fistulizing Crohn's disease), assuming patients have had inadequate responses to conventional therapy. It is not approved for the treatment of GVHD.

This is a Phase I pharmacokinetic study that is coordinated by the Pediatric Blood and Marrow Transplant Consortium (PBMTC). The study will be conducted in the Blood and Marrow Transplantation (BMT) program at Children's Healthcare of Atlanta - Egleston, Emory University Department of Pediatrics. The goal is to enroll 1 - 2 patients on this study; accrual will be via the BMT program. Eligible patients must be less than 18 years of age.

Patients with newly diagnosed acute GVHD will be able to participate in the study. Patients will receive a single dose of infliximab in the clinic. Since this is a Phase I study, the patients will have blood samples drawn to measure the pharmacokinetics of the drug. A total of 16 blood samples will be drawn over 84 days. The samples will be labeled with a code, processed, frozen, and then sent in a batch to the PBMTC designated laboratory for testing. Patients will continue on any drugs they were getting for the prevention of GVHD. Additional doses of infliximab may be given. This decision will be based on the results of the blood testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received corticosteroids at >= 2 mg/kg/day for a minimum of 72 hours prior to study entry.
* Overall clinical grade II-IV acute GVHD (aGVHD) with intestinal involvement with biopsy of at least one site "consistent with" aGVHD. Acute GVHD is defined in this study as occurring within 100 days after transplant.
* Men and women of childbearing potential must use adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) for the duration of the study and should continue such precautions for 6 months after receiving the study drug infusion.
* Parent(s)/legal guardian must give informed consent

Exclusion Criteria:

* Patients with uncontrolled infection(s), i.e. documented bacterial, viral or fungal infection within 72 hours prior to study entry. Neither continuation of antibiotics for a controlled infection nor prophylactic/empiric antibiotics warrant exclusion.
* Patients with any one of the following opportunistic infections documented within 8 weeks prior to study entry are excluded: cytomegalovirus disease, pneumocystis carinii, aspergillosis, histoplasmosis, atypical mycobacterium infection or other pathogenic molds/fungi.
* Serum creatinine > 1.5 mg/dl at study entry.
* Women who are pregnant, nursing, or planning pregnancy within 6 months following study drug infusion.
* Use of any investigational drug for the treatment of acute GVHD within 14 days prior to study entry. An investigational drug is defined as one that is being given on study, requiring informed consent.
* Use of ATG or similar product within 14 days prior to study entry requires study chair approval. Judgment will be based on ATG dosing and timing.
* Previous administration of infliximab.
* Any allergy to murine products.
* Documented HIV infection.
* Patients with grade IV renal, hepatic, pulmonary, or neurologic toxicity by National Cancer Institute (NCI) Common Toxicity Criteria (CTC).
* Patients with any history of congestive heart failure, defined as cardiac dysfunction requiring inotropic support other than dopamine at <= 5 mcg/kg/minute.
* Peripheral neuropathy or any demyelinating disease, greater than CTC grade 1.
* Presence of a transplanted solid organ (with the exception of a corneal transplant > 3 months prior to screening).
* Any prior history of tuberculosis (TB). Patients with a recent close contact with an individual with active TB are excluded. Patients with a household member who has a history of pulmonary TB should have a thorough evaluation for TB prior to study enrolment as recommended by a local infectious disease specialist or by guidelines on TB screening published by the United States (US) Federal Centers for Disease Control and Prevention (CDC).

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Dates: Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Sleight, M.D., Study Chair — Yale University
Locations (1):
- Children's Healthcare of Atlanta/Emory University, Atlanta, Georgia, United States